CLINICAL TRIAL: NCT01055366
Title: ELAZOP Switching Study in Korea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RM-09-06
Record Dates: First submitted 2010-01-22; First posted 2010-01-25 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-05

CONDITIONS: Open Angle Glaucoma
Keywords: Open angle glaucoma; OAG; Elazop; Azarga; Brinzolamide/Timolol combination
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Azarga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Elazop (Azarga) (Experimental): Elazop Treatment arm
  Interventions: Drug: Elazop (Azarga)

INTERVENTIONS:
Drug: Elazop (Azarga) — Administer one drop of ELAZOP in treated eye(s) twice a day for up to 12 weeks

SUMMARY:
The purpose of this study is to assess the safety and efficacy of switching to ELAZOP from prior pharmacotherapy in patients with open-angled glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Clinical diagnosis of ocular hypertension, primary open-angle or pigment dispersion glaucoma in both eyes.
* Must be on a stable regimen of Intraocular Pressure (IOP) lowering medication (i.e., either a single therapeutic agent or two separate ocular hypotensive agents) for at least one month prior to the Screening Visit.
* Must have IOP considered to be safe (in the opinion of the investigator), in both eyes, in such a way that should assure clinical stability of vision and the optic nerve throughout the study period.
* Must be willing to discontinue the use of all other ocular hypotensive medications prior to receiving the study medication for the entire course of the study.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Known medical history of allergy, hypersensitivity, or poor tolerance to any component of the preparations to be used in the study that is deemed clinically significant in the opinion of the Principal Investigator.
* Intraocular conventional surgery or laser surgery in either eye less than three months prior to the Screening visit.
* History of ocular herpes simplex.
* Pregnant or lactating.
* Participation in any other investigational study within 30 days of Screening visit.
* Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2010-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Mean Intraocular Pressure (IOP) change from baseline at final visit. | 12 weeks after treatment

CONTACTS AND LOCATIONS:
Locations (10):
- South Korea (10):
  - Youngnam Univ. Hospital, Daegu, Daegu
  - Seoul National University Bundang Hospital, Sungnam, Gyounggi
  - Seoul National University Hospital, Seoul
  - Yonsei University Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Yonsei University Kangnam Severance Hospital, Seoul
  - Seoul St. Mary's Hospital, The Catholic University of Korea, Seoul
  - Asan Medical Center, Seoul
  - Kim's Eye Hospital, Seoul
  - St. Mary's Hospital, The Catholic University of Korea, Seoul